CLINICAL TRIAL: NCT06915818
Title: GI Windows Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating Ileo-colic and Colo-colonic Anastomoses in Patients Undergoing Surgical Procedures
Brief Title: Flexagon Plus OTOLoc Colon Anastomosis in Patients Undergoing Surgery
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 25-003
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colon Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Study Group: Prospective Evaluation of Flexagon SFM Device with OTOLoc (Experimental): This is a multicenter, single-arm study in which clinical outcomes are prospectively evaluated for subjects undergoing ileo-colic and colo-colonic anastomosis using the Flexagon SFM Device with OTOLoc.
  Interventions: Device: Ileo-colic and colo-colonic Anastomosis with Flexagon SFM and OTOLoc

INTERVENTIONS:
Device: Ileo-colic and colo-colonic Anastomosis with Flexagon SFM and OTOLoc — This study will investigate two types of intervention: ileo-colic and colo-colonic anastomosis creation in subjects undergoing colon surgery. Flexagon SFMs and OTOLoc devices will be delivered laparoscopically and/or endoscopically into a portion of either the ileum or the colon that are intended to be anastomosed. An OTOLoc device will be deployed into the ileum/colon wall to provide access for the deployment of a Flexagon SFM into the bowel. The process is repeated at an intended section of colon. Once deployed, the Flexagon SFMs are approximated and positioned, after which the SFMs are couple together to form the anastomosis, with the OTOLoc devices allowing fluidic communication between the two lumens until the anastomosis is fully formed.

SUMMARY:
The primary objective of this trial is to investigate the safety and effectiveness of the Flexagon SFM system plus OTOLoc when used to create a Ileo-colic and Colo-colonic anastomoses in participants undergoing colon surgery.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical study to evaluate the GI Windows Flexagon Self Forming Magnet Anastomosis plus OTOLoc for creating Ileo-colic and Colo-colonic anastomoses in participants undergoing colon surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22 years or older at screening
2. Candidate for surgery requiring Right Hemicolectomy or Sigmoid / Low Anterior resection (with anastomosis above the peritoneal reflection) with cardiac/medical clearance for surgery
3. Able to understand and sign informed consent document
4. American Society of Anesthesiologists (ASA) score < IV at time of procedure
5. All cancer patients must have completed chemotherapy ≥2 months prior to procedure
6. Lives, and intends to remain, within a 300 kilometers radius of study center for the duration of the study
7. Able to refrain from smoking during study follow-up period

Exclusion Criteria:

1. Known or suspected allergy to silicone, nickel, titanium or Nitinol
2. BMI > 55 kg/m2
3. Uncontrolled diabetes (defined as HbA1c >10%)
4. Congenital or acquired anomalies of the GI tract, including atresia or malrotation that would inhibit passing of SFM magnet
5. Diagnosed with obstructed or perforated colon cancer
6. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy that may suggest difficulty during endoscopic delivery of magnets
7. Any previous major surgery on the stomach, duodenum, hepatobiliary tree, pancreas, Whipple or right colon
8. History of recurrent small bowel obstructions.
9. Coagulation deficiency not normalized by medical treatment or platelet count <50,000/µL
10. Known moderate to severe renal disease (eGFR < 44 milliliters per minute per 1.73m2) or ongoing dialysis
11. Hyperkalemia / hypercoagulability or prior Venus Thromboembolism / Pulmonary Embolism
12. Immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e., 20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents
13. Congestive heart failure with ejection fraction <35% or clinically significant arrhythmia (any rhythm disturbances except sinus tachycardia, sinus bradycardia or a sinus rhythm with premature atrial or ventricular complexes)
14. Decompensated chronic obstructive lung disease
15. Active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound.
16. Contraindication to general anesthesia
17. Breast-feeding, pregnant, or planning on becoming pregnant during the follow-up period
18. Currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent
19. Contraindication to general anesthesia
20. Participant is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successful Anastomosis Creation without the Need for Reoperation | 30 Days
  The study's primary endpoint (patient success) is defined as successful anastomosis created with the Flexagon SFM without placement procedure, device or target anastomosis-related reoperation through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, Principal Investigator — Mohak Hitech Specialty Hospital; Vinod Dhakkad, MD, Principal Investigator — Mohak Hitech Specialty Hospital; Pablo Marin, MD, Principal Investigator — Clinica Colonial Hospital
Locations (2):
- Clinica Colonial Hospital, Santiago, Huechuraba, Región Metropolitana, Chile
- Mohak Hitech Specialty Hospital, Indore, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.